CLINICAL TRIAL: NCT06905821
Title: The Effect of Antenatal Education Based on Transformative Learning Theory on Traumatic Birth Perception, Fear of Birth, and Birth Readiness in Pregnant Women: a Randomized Controlled Trial
Brief Title: Effects of Antenatal Education on Birth Perception, Fear, and Readiness
Acronym: EA-BPFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Şahika ŞİMŞEK ÇETİNKAYA, Head of Midwifery, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-KAEK-41
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-06

CONDITIONS: Childbirth; Fear
Keywords: Transformative Learning; pregnancy; fear; trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transformational Learning-Based Antenatal Education Group (Experimental): This group will receive antenatal education based on transformational learning theory. The program aims to reduce birth fear and traumatic birth perception by providing participants with targeted information and strategies. Participants will gain knowledge and coping mechanisms to manage pain, stress, and anxiety during labor. The education will focus on raising awareness about the birth process, promoting psychological preparedness, and supporting post-birth recovery, all aimed at enhancing overall birth experience and well-being
  Interventions: Behavioral: Transformational Learning-Based Antenatal Education Program
- Standard Antenatal Care Group (No Intervention): This group will receive standard antenatal care, which includes routine check-ups and general health education related to pregnancy. Participants will not receive the transformational learning-based antenatal education or any specific intervention related to birth fear or traumatic birth perception. The standard care focuses on general information about the physiological process of pregnancy and labor but does not address psychological preparedness or provide strategies for managing birth-related anxiety or fear.

INTERVENTIONS:
Behavioral: Transformational Learning-Based Antenatal Education Program — The Transformational Learning-Based Antenatal Education Program helps pregnant women reduce birth-related anxiety and fear by utilizing transformational learning theory. Unlike traditional antenatal education, it emphasizes psychological preparedness, focusing on emotional well-being and coping strategies. The program includes interactive learning, group discussions, and self-reflection to engage participants actively. This approach aims to boost women's confidence and reduce stress as they approach labor and delivery.
  Arms: Transformational Learning-Based Antenatal Education Group

SUMMARY:
Birth is a multi-dimensional and unique experience for every woman, and it is influenced by a woman's social life. Fear of childbirth is a common issue that affects women's health and well-being before, during, and after pregnancy. The thought that childbirth will be painful triggers fear of childbirth. Fear of childbirth is closely related to the perception of traumatic birth. Antenatal education is important in coping with childbirth pain and traumatic birth pain, but the aim of adult education is not just to inform, but also to change individuals' perspectives on events. The transformative learning theory is a model used to change individuals' perspectives on events. The aim of this study was to investigate the effect of antenatal education based on the transformative learning theory on traumatic birth perception, fear of childbirth, and birth preparedness in pregnant women. The study was conducted as a randomized controlled trial with 54 participants. Data collection forms included a personal information form, the Traumatic Birth Perception Scale, the Prenatal Self-Assessment Scale, and the Wijma Birth Expectancy/Experience Scale. The Statistical Package for the Social Sciences 23.0 (Chicago, Illinois) version was used for data analysis. Histogram and Q-Q plots, and the Shapiro-Wilk test were used to assess the normality of the data distribution. Descriptive data regarding women's demographic characteristics were analyzed using frequencies, percentages, and mean values. Differences in demographic characteristics between groups were examined using the independent sample t-test, Mann-Whitney U test, and Chi-square test. Pre-test and post-test scores of the groups were analyzed using the independent sample t-test. A significance level of p<0.05 was accepted.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 20-35
* Be in the 30-32 weeks of gestation
* Be a primigravida
* Have at least basic literacy skills

Exclusion Criteria:

* Have any chronic diseases
* Have any psychiatric disorders
* Be a high-risk pregnancy
* Have any communication problems
* Have communication issues

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Perception of Traumatic Birth | Baseline: Week 30 of pregnancy (pre test); An average of 3 weeks (post test)
  This will be assessed using the Traumatic Birth Perception Scale.The scale, developed by Yalnız et al. (2016), is called the Traumatic Birth Perception Scale. It is designed to assess the traumatic birth perception levels of women of reproductive age. It consists of 13 items that encompass the thoughts and emotions, such as anxiety, fear, and concern, that a woman experiences when thinking about childbirth. For each item, respondents rate their feelings on a scale from 0 ("no fear") to 10 ("extreme fear"). The total average score indicates the level of traumatic birth perception. The lowest and highest possible scores on the scale are 0 and 130, respectively. As the score increases, it reflects a higher perception of traumatic birth. The score ranges are as follows: 0-26 indicates very low, 27-52 low, 53-78 moderate, 79-104 high, and 105-130 indicates very high levels of traumatic birth perception. The Cronbach's alpha reliability coefficient of the scale is 0.89.

SECONDARY OUTCOMES:
Childbirth Readiness | Baseline: Week 30 of pregnancy (pre test); An average of 3 weeks (post test)
  The Childbirth Readiness Subscale (PKDÖ-DHOÖ) was developed by Lederman in 1979 to assess women's adaptation to motherhood during the prenatal period. The scale, consisting of 79 items and using a 4-point Likert-type scale, was validated and tested for reliability in Turkey by Beydağ and Mete (2008). The scale includes 7 subscales: thoughts about the health of oneself and the baby, acceptance of pregnancy, acceptance of the maternal role, childbirth readiness, fear of childbirth, relationship with the mother, and relationship with the spouse. These subscales can be used independently. The general Cronbach's alpha for the Turkish version of the scale is 0.81, and the internal consistency reliability coefficients for the subgroups range from 0.72 to 0.85 (Beydağ & Mete, 2008). Scores on the scale range from 10 to 40. The Cronbach's alpha value for the Childbirth Readiness Subscale (DHOÖ) is 0.72. As the score increases, it indicates a lower level of readiness for childbirth.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu, Kastamonu, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No